CLINICAL TRIAL: NCT06020248
Title: Melanin and Dermal Uptake of Thirdhand Cigarette Smoke
Acronym: THS05
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-37861
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Thirdhand tobacco smoke; Dermal; Exposure; Tobacco Smoke Pollution; Melanin; Nicotine

STUDY DESIGN:
Intervention Model Description: Dermal uptake, metabolism and excretion of nicotine in participants with high and low levels of dermal melanin will be compared.
Masking Description: Smoke exposure is impossible to mask and team is too small to mask data analysis until later stages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low melanin (Experimental): Individuals with skin reflectance scores below 150 using the Mexameter 18 instrument.
  Interventions: Other: Wear clothing that has been exposed to cigarette smoke for 3 hours.
- High melanin (Experimental): Individuals with skin reflectance scores above 249 using the Mexameter 18 instrument
  Interventions: Other: Wear clothing that has been exposed to cigarette smoke for 3 hours.

INTERVENTIONS:
Other: Wear clothing that has been exposed to cigarette smoke for 3 hours. — Cotton clothing is exposed to smoke from Marlboro Red (hard pack) cigarettes at 1-1.2 mg/m3 repeatedly, until total exposure equals 3 grams total particulate material. When tested after exposure, the clothing typically contained 59.15 +/- 18 µg nicotine and 42 +/- 24 ng NNK per gram. The mass of the clothing varies by size, but the average combination of pants and shirt contains 32 mgs nicotine and 23 µg NNK.

SUMMARY:
This is a pilot study of the effects of dermal melanin on dermal uptake and retention of nicotine. The initial hypothesis is that higher levels of dermal melanin will correlate with lower uptake and longer retention of nicotine in the skin and body.

DETAILED DESCRIPTION:
This is an interventional pharmacokinetic study comparing the uptake and metabolism of nicotine from smoke-exposed clothing in people with low high levels of dermal melanin and people with high levels of dermal melanin. The study will measure nicotine and metabolites of nicotine in the blood during exposure and in urine for 10 days after exposure.

ELIGIBILITY:
Inclusion Criteria:

* Adult nonsmoker
* Aged 18-50
* Skin reflectance scores below 150 or above 249 using the Mexameter 18 instrument
* Healthy on the basis of medical history
* Systolic blood pressure <150
* Diastolic blood pressure <100
* C-reactive protein <3.1 mg/ml
* Liver function (AST and ALT) in normal ranges
* kidney function (BUN) in normal ranges
* LDL<131
* Blood glucose <110
* Not exposed to tobacco SHS.

Exclusion Criteria:

* Dermal skin reflectance score between 150 and 249, as measured by the Mexameter 18 instrument.
* Positive SARS-CoV-2 antibody test
* Age 18 < or > 50
* Physician diagnosis of asthma, heart disease, hypertension, thyroid disease, diabetes, renal or liver impairment or glaucoma.
* Unstable psychiatric condition (such as current major depression, history of schizophrenia or bipolar disorder) or current use of more than two psychiatric medications
* Systolic blood pressure greater than or equal to 150
* Diastolic blood pressure greater than or equal to 100
* Blood glucose greater than or equal to 110
* LDL greater than or equal to130
* Pregnancy or breastfeeding (by urine hCG and/or history)
* Alcohol or illicit drug dependence within the past 5 years
* BMI > 35 and < 18
* Current illicit drug use (by history or urine test)
* More than 1 pack year smoking history
* Ever a daily marijuana smoker
* Smoked anything within the last 3 months
* Unable to hold allergy or other OTC medicines
* Occupational exposure to smoke, dusts OR fumes
* Concurrent participation in another clinical trial
* Unable to communicate in English
* No social security number

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in blood concentrations of nicotine | Baseline and 3 hours
  The study will measure concentration of nicotine in the blood before and after the dermal exposure to nicotine.
Total combined urinary concentrations of the nicotine metabolites cotinine and 3-hydroxycotinine | First void, collected for 10 days
  The study will measure urinary metabolites of nicotine in the first void of the day for 10 days after exposure and sum the total mass of metabolites.

SECONDARY OUTCOMES:
Urinary concentration of the NNK metabolite NNAL | First void, collected for 10 days
  The study will measure urinary metabolites of NNK in the first void of the day for 10 days after exposure and sum the total mass of metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Suzaynn F Schick, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No